CLINICAL TRIAL: NCT07053878
Title: Impact of Non-Surgical Periodontal Therapy on Awake and Sleep Bruxism in Patients With Stage III-IV Periodontitis
Brief Title: Changes in Bruxism Activity After Periodontal Treatment in Patients With Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Nicola Discepoli, Associate Professor, University of Siena
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PB002
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Periodontitis; Bruxism; Sleep Bruxism; Awake Bruxism
MeSH Terms: conditions — Periodontitis; Bruxism; Sleep Bruxism

STUDY DESIGN:
Intervention Model Description: Two-group, non-randomized controlled pre-post study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodontitis Group (Experimental): Participants with Stage III or IV periodontitis will receive full non-surgical periodontal therapy (step 1 and step 2), along with standardized oral hygiene instructions and motivation. Bruxism activity and periodontal status will be assessed at baseline and after three months.
  Interventions: Procedure: Non-Surgical Periodontal Therapy (Step 1 & 2)
- Healthy Control Group (Active Comparator): Periodontally healthy participants will receive supragingival plaque removal and polishing, along with standardized oral hygiene instructions and motivation. Bruxism activity and periodontal status will be assessed at baseline and after three months.
  Interventions: Procedure: Supragingival Plaque Removal and Polishing

INTERVENTIONS:
Procedure: Non-Surgical Periodontal Therapy (Step 1 & 2) — Comprehensive supra- and sub-gingival instrumentation (scaling, root planing, ultrasonic and manual instruments), following EFP step-1 and step-2 protocols. Includes individualized oral-hygiene instruction and motivation.
  Arms: Periodontitis Group
Procedure: Supragingival Plaque Removal and Polishing — Professional supragingival scaling with ultrasonic tips plus rubber-cup polishing in a single session. Includes the same individualized oral-hygiene instruction and motivation provided to the experimental group.
  Arms: Healthy Control Group

SUMMARY:
This controlled pre-post study evaluates the effect of non-surgical periodontal therapy on awake and sleep bruxism in patients with Stage III and IV periodontitis. Bruxism activity and periodontal status will be assessed at baseline and three months after treatment.

DETAILED DESCRIPTION:
This is a non-randomized controlled pre-post clinical study designed to investigate the impact of periodontal treatment on awake and sleep bruxism in individuals with advanced periodontitis. Two groups will be included: a periodontitis group undergoing full non-surgical periodontal therapy (step 1 and 2), and a healthy control group receiving supragingival plaque removal and polishing. All participants will receive standardized oral hygiene instructions and motivation. Bruxism activity will be recorded using portable electromyography (EMG) devices at baseline and after three months, evaluating both sleep and awake bruxism through Bruxism Work Index (BWI) and Bruxism Time Index (BTI). Clinical periodontal parameters will also be collected at both time points to assess potential correlations with bruxism variation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25 and 50 years
* Good general health (ASA I or II)
* Signed informed consent
* Willingness to attend all study visits and follow instructions
* For periodontitis group: diagnosis of Stage III or IV periodontitis according to the 2017 classification
* For healthy control group: no clinical signs of periodontitis

Exclusion Criteria:

* Systemic diseases or medications affecting the periodontium (e.g., diabetes, immunosuppressants)
* Antibiotic or anti-inflammatory therapy within the last 3 months
* Periodontal treatment in the last 6 months
* Smoking more than 10 cigarettes/day
* Use of occlusal splints or bruxism-targeted therapy in the past 6 months
* Pregnancy or lactation
* Any condition impairing the ability to cooperate or comply with the study protocol

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-06-27 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Bruxism Episodes | Baseline and 3 months
  Number of bruxism events measured using portable electromyographic (EMG) devices, at baseline and after periodontal/prophylactic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Discepoli, DDS, PhD, Principal Investigator — Department of Medical Biotechnologies, University of Siena
Locations (1):
- AOUS, Siena, Italy